CLINICAL TRIAL: NCT06872307
Title: Intervention to Enhance Prep Persistence Among African American Men Who Have Sex with Men
Brief Title: Intervention to Enhance PrEP Persistence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Whitman-Walker Institute (Other Government); Rhode Island Public Health Institute (Unknown); University of Mississippi Medical Center (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amy Nunn, Professor of Public Health and Medicine at Brown University; Executive Director of the Rhode Island Public Health Institute, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000087; 1R01MH131475-01A1 (NIH)
Record Dates: First submitted 2024-10-17; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-10

CONDITIONS: HIV Prevention; HIV Infection Primary
Keywords: pre-exposure prophylaxis

STUDY DESIGN:
Intervention Model Description: All eligible participants will be randomly assigned to either the RAMP-It-Up intervention or control condition with a 1:1 ratio stratified by study site. Randomization will occur immediately following participants' completion of baseline activities. Block randomization (with random block size of 4 or 6) will be used to achieve a nearly balanced number of participants in the intervention and control arms at any given time point at each site.121 Each study site will receive a list of random treatment assignments generated by a statistical algorithm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Control Arm) (No Intervention): Standard of care (access to a financial advocate and clinical staff to support, facilitate, and assist in linkage to the established PrEP clinic at study sites and to facilitate initiation of, and obtaining, PrEP medications)
- RAMP-It-Up intervention (Experimental): The RAMP-It-Up intervention focuses on personalized navigation informed by strengths-based case management. RAMP-It-Up consists of a brief in-person patient navigation session, ongoing bidirectional communication as needed, short (10-minute) phone or text message check-ins with the navigator, strengths-based case management strategies to overcome barriers, optional daily medication text reminders, transportation assistance to clinical visits as needed, and monthly calls to patients' pharmacies to assess prescription pick-up, allowing the navigator to provide real-time support in addressing barriers to PrEP initiation, adherence, and retention in care.
  Interventions: Behavioral: RAMP-It-Up Initiation, Adherence, and Retention Intervention

INTERVENTIONS:
Behavioral: RAMP-It-Up Initiation, Adherence, and Retention Intervention — The intervention arm will receive facilitated strengths-based case management (SBCM)-delivered by trained interventionists-to help navigate the PrEP medical care system and support the participant and health care staff in meeting the challenges faced with obtaining PrEP medication (e.g., overcoming insurance barriers or barriers with co-pays). This also includes facilitated integration into the PrEP clinic and obtaining monthly PrEP prescription refills
  Arms: RAMP-It-Up intervention

SUMMARY:
The investigators will conduct a fully powered randomized controlled trial (RCT) to test the effect of a patient navigation intervention for Black/African American (B/AA) men who have sex with men (MSM) on PrEP initiation, adherence and retention in care. B/AA men who have sex with men (MSM) are disproportionately impacted by the HIV/AIDS epidemic in the United States. Pre-exposure prophylaxis (PrEP), a once daily medication, can dramatically reduce HIV acquisition risk. However, social and structural barriers have contributed to suboptimal PrEP initiation, adherence, and retention in care among B/AA MSM. Our prior NIH-funded pilot study (R34MH109371; MPI: Nunn, Chan, Mena) developed and evaluated an Intervention to Retain and Adhere MSM in PrEP (RAMP-IT-UP), a brief strengths-based patient navigation program to enhance PrEP care outcomes among young B/AA MSM. The intervention was found to be highly acceptable among B/AA MSM and demonstrated preliminary effectiveness. Compared to control participants, RAMP-IT-UP participants were statistically more likely to initiate PrEP and adhere to PrEP based on pharmacy fill data and PrEP blood levels. Additionally, RAMP-IT-UP participants were more likely to be retained in PrEP care at the 3-month and 6-month clinical visits. Specific Aim #1 of this study will conduct a fully powered randomized controlled trial (RCT to estimate the effectiveness of RAMP-IT-UP in improving PrEP adherence and care outcomes among B/AA MSM in real-world community health center settings (CHCs). Specific Aim #2 will estimate the cost-effectiveness of RAMP-IT-UP among B/AA MSM attending CHCs compared to standard of care. The investigators will also determine the cost-effectiveness of differing levels of intensity of navigation services to prevent HIV based on data collected in Specific Aim #1. Our goal is to develop a cost-effective intervention that enhances PrEP care outcomes and reduces HIV incidence for B/AA MSM which will be relevant for CHCs across the US. The long-term goal of this work is to decrease HIV incidence among B/AA MSM, which aligns with federal Ending the HIV Epidemic and National HIV/AIDS Strategy goals. This application is led by an experienced team of investigators with a proven track record conducting HIV, PrEP and disparities research in real-world clinical settings.

DETAILED DESCRIPTION:
Black/African American (B/AA) gay, bisexual, and other men who have sex with men (MSM) are at high risk for HIV acquisition in the United States (US). Although B/AA MSM account for less than 1% of the US population, they comprise 26% of new HIV infections. An estimated 41% of B/AA MSM acquire HIV during their lifetimes. HIV pre-exposure prophylaxis (PrEP) can dramatically reduce HIV incidence for B/AA MSM.

B/AA MSM have poorer outcomes at every stage of the PrEP care continuum. B/AA MSM are less likely to initiate PrEP, and be retained in care than non-Hispanic White MSM. PrEP care outcomes among B/AA MSM are influenced by complex social and structural factors, such as difficulty accessing culturally congruent healthcare services, insufficient health insurance, high out-of-pocket costs, and stigma associated with PrEP, sexual orientation, and HIV. The US Ending the HIV Epidemic (EtHE) initiative and the National HIV/AIDS Strategy call for expanding PrEP to B/AA MSM at community health centers (CHCs), but few interventions exist to overcome barriers and improve PrEP care outcomes in this setting. Moreover, access to PrEP navigation services in real-world settings is uneven. While some clinics offer PrEP navigation services, there is no standard or scientific consensus about how to enhance PrEP adherence and retention in care for B/AA MSM. There is also a lack of data on the degree of intensity and time for navigation services to achieve optimal PrEP outcomes for this population.

The investigator's NIH-funded pilot randomized controlled trial (RCT) (R34MH109371; MPI: Nunn, Chan, Mena) developed and evaluated the Retain and Adhere MSM on PrEP Intervention (RAMP-IT-UP), a strengths-based patient navigation program to enhance PrEP care outcomes among B/AA MSM at a CHC in Jackson, Mississippi. RAMP-IT-UP included one 60-minute personalized patient navigation session, bidirectional communication, scheduled short (10-minute) phone check-ins with navigators, tailored strengths-based strategies to overcome barriers, optional tailored daily medication reminders via text message, and transportation assistance as needed. RAMP-IT-UP also included monthly calls to patients' pharmacies to assess prescription pick-ups, allowing the navigator to connect with patients in a timely manner to understand why a PrEP prescription was not filled. RAMP-IT-UP provides real-time support to overcome social, structural and clinical barriers to PrEP initiation, retention, and adherence and was highly acceptable among B/AA MSM. Compared to control participants, RAMP-It-Up participants were much more likely to initiate PrEP (93% vs. 63%, p=0.01) and to adhere to PrEP based on pharmacy fill data (70% vs. 23%, p<0.01) and 3-month drug levels (83% vs. 50%, p=0.20). Additionally, RAMP-It-Up participants were more likely to be retained in PrEP care at 3-month (70% vs. 43%, p=0.05) and 6-month (37% vs. 27%, p=0.42) PrEP visits.

The objectives of the proposed study are to conduct a fully multi-site RCT to determine the effectiveness and cost-effectiveness of RAMP-It-Up for improving PrEP care outcomes among B/AA MSM in real-world CHC settings. The long-term goal of this work is to decrease HIV incidence among B/AA MSM, which aligns with EtHE and National HIV/AIDS Strategy goals. The investigators propose the following specific aims:

Specific Aim #1: Conduct a fully powered RCT to estimate the effectiveness of RAMP-It-Up among B/AA MSM attending CHCs. The investigators will enroll n=300 B/AA MSM who intend to initiate daily oral PrEP at CHCs in three US urban centers (N=100 each site): Jackson, Mississippi; Washington, District of Columbia; and Providence, Rhode Island. Block randomization will be used to randomize participants at each site to either RAMP-IT-UP or an attention-matched information/referral control condition (enhanced treatment-as usual [ETAU]). Quantitative research assessments will be conducted at baseline and 3-, 6-, 9-, and 12-months post-baseline. The primary outcome will be PrEP adherence, given that adherence is the definitive marker associated with protection from HIV infection. The investigators will measure adherence with pharmacy refill data and validate pharmacy refill data with PrEP drug levels. Secondary analyses will evaluate PrEP initiation and retention in care at clinical visits. The investigators hypothesize that, compared to ETAU, RAMP-It-Up will significantly improve PrEP initiation, adherence, and retention in care outcomes.

Specific Aim #2: Estimate the cost-effectiveness of RAMP-It-Up among B/AA MSM attending CHCs compared to ETAU. The investigators will employ intervention costing methods to evaluate costs of delivering RAMP-It-Up based on a comprehensive suite of tailored navigation services compared to ETAU. The investigators will then use a Markov state-transition model to estimate the cost-effectiveness of RAMP-It-Up compared to ETAU, in terms of cost-per-person initiating PrEP, adhering to PrEP, and being retained in PrEP care. The investigators will also determine the cost-effectiveness of differing levels of intensity of navigation services to prevent HIV based on data collected in Specific Aim #1. The ultimate goal is to develop a cost-effective intervention that enhances PrEP care outcomes and reduces HIV incidence among B/AA MSM that will be relevant for CHCs. This study is led by a highly successful research team with a long-standing history of collaboration on PrEP implementation studies in real-world settings. This proposal aligns with EtHE and National HIV/AIDS Strategy goals of scaling PrEP in real-world settings in geographic hotspots, with a focus on B/AA MSM.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Assigned male sex at birth
* Identify as Black/African American
* Report at least one male sex partner in the past 12 months
* Meet the CDC eligibility criteria for PrEP
* Have not taken PrEP for at least 30 days
* Are HIV-negative based on antibody testing at the time of enrollment
* Understand and speak English
* Able to provide informed consent
* Agree to authorize study access to their EHR and pharmacy fill data. Eligible patients who are interested in participating will be consented and enrolled into the study.

Exclusion Criteria:

* Under the age of 18
* Assigned female sex at birth
* Does not identify as Black/African American
* Has not had a male sex partner in the past 12 months
* Does not meet CDC eligibility criteria for PrEP
* Has taken PrEP within the last 30 days
* HIV-positive or inconclusive HIV status based on antibody testing at the time of enrollment
* Does not understand or speak English
* Unable to provide informed consent
* Does not agree to authorize study access to their EHR and pharmacy fill data.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
PrEP Adherence - Pharmacy Fill Data | 3 and 12 Month Follow Ups
  The primary outcome will be PrEP adherence, given adherence is the definitive marker associated with protection from HIV infection. Adherence will be measured using pharmacy fill data in order to determine whether participants have picked up their prescription on a monthly basis.
PrEP Adherence - Drug Levels | 3 and 12 Month Follow Ups
  The primary outcome will be PrEP adherence, given adherence is the definitive marker associated with protection from HIV infection. Adherence will be assessed by dried blood spot sampling for PrEP drug levels.

SECONDARY OUTCOMES:
PrEP Initiation | 3 and 12 Month Follow Ups
  PrEP initiation will be measured as a secondary outcomes. This will be assessed by whether participants successfully obtained a PrEP prescription.
PrEP Retention in Care | 3 and 12 Month Follow Ups
  PrEP retention in care will be measured as a secondary outcome. Retention in care will be quantified by the number of PrEP clinical visits attended or missed in the 12 months after initiation.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Whitman Walker Health, Washington D.C., District of Columbia
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Rhode Island Public Health Institute, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No